CLINICAL TRIAL: NCT03393910
Title: The Improvement Of Pelvic Exams for Patients With Chronic Vulvovaginal Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Rebecca Rinko, Dr. Rebecca Rinko, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DrexelU
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational (No Intervention): Normal pelvic exam exposures: External exam followed by speculum exam, followed by bimanual exam
- Experimental Pelvic Exam (Active Comparator): Changing the order of the pelvic exam Intervention: External exam, bimanual exam,speculum exam
  Interventions: Diagnostic Test: Experimental Pelvic Exam

INTERVENTIONS:
Diagnostic Test: Experimental Pelvic Exam — The pelvic exam will be completed in the following order: external, speculum, bimanual exam in the "standard" group. In the Experimental group the pelvic exam will be done with external xam, bimanual exam then speculum exam.
  Arms: Experimental Pelvic Exam

SUMMARY:
The purpose of this study is to investigate patients self-reported comfort levels during each section of the pelvic exam.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to investigate the sequence in which physicians perform the pelvic exam, describe and compare self-reported comfort during each section of the pelvic exam and how comfort during the examinations related to quality of life, self-esteem, and sexual function in English speaking females at least 18 years of age with chronic vulvovaginal conditions.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking Are able to read and write English Are utilizing outpatient services and being seen for a first appointment at an outpatient Vulvodynia Center

Exclusion Criteria:

* Non English Speaking
* Patients who cannot read or write
* Those who are pregnant
* Those who do not have a chronic vulvovaginal condition
* Patients other than "new" patients
* Patients who would not otherwise need a speculum exam

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score: A change of 13mm | Within 1 hour of the exam
  ale from 0-10, measured in mm. A change from baseline of 13mm is considered a significant change

SECONDARY OUTCOMES:
Wellbeing quality of life score: Range 0-4 | Within 1 hour of the exam
  High wellbeing 2.504.0, Low Wellbeing 1.5-2.4, and very low wellbeing 0-1.4
Rosenberg Self-esteem Score: Scale 10-40 | Within 1 hour of the exam
  Higher numbers indicate higher self-esteem
Female Sexual Function Index-19 | Within 1 hour of the exam
  Score of less than 26.55 indicates sexual dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel Ob/Gyn, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams AA, Williams M. A guide to performing pelvic speculum exams: a patient-centered approach to reducing iatrogenic effects. Teach Learn Med. 2013;25(4):383-91. doi: 10.1080/10401334.2013.827969. PMID 24112210
- [Background] Hilden M, Sidenius K, Langhoff-Roos J, Wijma B, Schei B. Women's experiences of the gynecologic examination: factors associated with discomfort. Acta Obstet Gynecol Scand. 2003 Nov;82(11):1030-6. doi: 10.1034/j.1600-0412.2003.00253.x. PMID 14616277
- [Background] Wijma B, Gullberg M, Kjessler B. Attitudes towards pelvic examination in a random sample of Swedish women. Acta Obstet Gynecol Scand. 1998 Apr;77(4):422-8. PMID 9598951
- [Background] Bernet R, Buddeberg C. [Physician-patient relations in gynecology: expectations and experiences of patients]. Gynakol Geburtshilfliche Rundsch. 1994;34(1):43-9. doi: 10.1159/000272333. German. PMID 8019173
- [Background] Daley AM, Cromwell PF. How to perform a pelvic exam for the sexually active adolescent. Nurse Pract. 2002 Sep;27(9):28, 31-2, 34, 37-9, 43; quiz 44-5. doi: 10.1097/00006205-200209000-00006. PMID 12352766
- [Background] Primrose RB. Taking the tension out of pelvic exams. Am J Nurs. 1984 Jan;84(1):72-4. No abstract available. PMID 6559035
- [Background] Nyirjesy P, Peyton C, Weitz MV, Mathew L, Culhane JF. Causes of chronic vaginitis: analysis of a prospective database of affected women. Obstet Gynecol. 2006 Nov;108(5):1185-91. doi: 10.1097/01.AOG.0000239103.67452.1a. PMID 17077241
- [Background] Goetsch MF, Lim JY, Caughey AB. Locating pain in breast cancer survivors experiencing dyspareunia: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1231-1236. doi: 10.1097/AOG.0000000000000283. PMID 24807329
- [Background] Dargie EE, Chamberlain SM, Pukall CF. Provoked Vestibulodynia: Diagnosis, Self-Reported Pain, and Presentation During Gynaecological Examinations. J Obstet Gynaecol Can. 2017 Mar;39(3):145-151. doi: 10.1016/j.jogc.2017.01.001. PMID 28343555
- [Background] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Background] Kelly AM. Does the clinically significant difference in visual analog scale pain scores vary with gender, age, or cause of pain? Acad Emerg Med. 1998 Nov;5(11):1086-90. doi: 10.1111/j.1553-2712.1998.tb02667.x. PMID 9835471
- [Background] Rowbotham MC. What is a "clinically meaningful" reduction in pain? Pain. 2001 Nov;94(2):131-132. doi: 10.1016/S0304-3959(01)00371-2. No abstract available. PMID 11690725
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton, NJ: Princeton University Press.
- [Background] Wiegel M, Meston C, Rosen R. The female sexual function index (FSFI): cross-validation and development of clinical cutoff scores. J Sex Marital Ther. 2005 Jan-Feb;31(1):1-20. doi: 10.1080/00926230590475206. PMID 15841702
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Derived] Rinko R, Spector C, Cook E, Mancenido B, Gracely EJ, Nyirjesy P. Sequence of Pelvic Examination Does Not Affect Patients With Baseline Vulvovaginal Syndromes: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Jan 1;27(1):e45-e51. doi: 10.1097/SPV.0000000000000791. PMID 32332423